CLINICAL TRIAL: NCT04141449
Title: A Multilevel Intervention (Potlako+) to Improve Timely Cancer Detection and Treatment
Brief Title: A Multilevel Intervention to Improve Timely Cancer Detection and Treatment Initiation
Acronym: Potlako+
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Botswana Harvard AIDS Institute Partnership (Other); Dana-Farber Cancer Institute (Other); National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Scott Lee Dryden-Peterson, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BHP0120; R01CA236546 (NIH)
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Neoplasms; Hiv; Cervical Cancer; Breast Cancer; HNSCC; Vulvar Cancer; Anal Cancer; Cancer Suspect
MeSH Terms: conditions — Neoplasms; Acquired Immunodeficiency Syndrome; Uterine Cervical Neoplasms; Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Vulvar Neoplasms; Anus Neoplasms

STUDY DESIGN:
Intervention Model Description: Paired, community-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potlako intervention (Experimental): * Provider oncology training focused on detection of cancer symptoms/signs and performance of appropriate diagnostic evaluation
  * Community-led cancer symptom awareness campaign to educate residents on methods and importance of early detection of cancer
  * Support/counselling call after initial clinician recognition that patient requires evaluation for possible cancer.
  * Cross-sectional community-facing activities partnered with longitudinal clinic-based targeted educational program
  * Remote phone/SMS-based cancer suspect navigation program to support and expedite evaluation for symptoms/signs of possible cancer.
  Interventions: Other: Potlako intervention
- Enhanced Care (Active Comparator): * Provider oncology training focused on detection of cancer symptoms/signs and performance of appropriate diagnostic evaluation.
  * Support/counselling call after initial clinician recognition that patient requires evaluation for possible cancer.
  Interventions: Other: Enhanced care

INTERVENTIONS:
Other: Potlako intervention — Combined provider, patient, and health system intervention to expedite cancer diagnosis and care.
  Arms: Potlako intervention
Other: Enhanced care — Provider education and limited patient counseling.
  Arms: Enhanced Care

SUMMARY:
This study evaluates whether the Potlako+ intervention of community education, clinical provider support, and patient navigation can improve access to cancer case for patients presenting with symptoms of cancer. Half of communities will receive the Potlako+ intervention, while the other communities will continue to receive standard programs.

DETAILED DESCRIPTION:
The Potlako+ trial is a pair-matched, community-randomized study involving 20 rural and peri-urban communities in Botswana (population ~190,100 with ~100,000 30 years or older). Communities will be randomized 1:1 to the Potlako+ intervention versus standard care. The goal of the intervention is to identify individuals with symptoms/signs suggestive of cancer and expedite diagnosis (and treatment).

The trial includes a community education component focused on cancer awareness and importance of early diagnosis and a patient navigation component that aims to expedite the diagnostic evaluation. Community education will be directed at approximately 50,000 community residents (30 years and older). We anticipate approximately 1500 cancer suspects will be identified by their clinic providers.

ELIGIBILITY:
1. Community members

   1. Inclusion Criteria:

      * Botswana citizen
      * Age 30 years or older
      * engaged in longitudinal care for chronic health problem
      * resident of study community
   2. Exclusion Criteria:

      * Involuntary incarceration
      * Educational messaging could interfere with clinical management or increase distress in the opinion or clinic or research staff
2. Cancer suspects

   1. Inclusion Criteria:

      * Botswana citizen
      * Age 30 years or older
      * resident of study community
      * Recorded as a cancer suspect by clinic staff
   2. Exclusion Criteria

      * Involuntary incarceration
      * Unable or unwilling to provide confirmation of informed consent
      * Already engaged in oncology care

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 874 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Duration of combined Appraisal and Help-seeking intervals | Baseline
  Number of days from patient symptom awareness to first clinic visit, among patients with moderate or high probability of cancer
Duration of Diagnostic interval | From date of first clinic visit to date of cancer diagnosis or diagnosis excluding cancer, up to 365 days
  Number of days from first clinic visit to cancer diagnosis or diagnosis excluding cancer, among patients with moderate or high probability of cancer
Duration of Pre-Treatment interval | From date of cancer diagnosis to date of cancer treatment up to 365 days
  Number of days from cancer diagnosis to cancer treatment
Proportion of patients treated with limited stage cancer | From date of cancer diagnosis to date of cancer treatment up to 365 days
  Among patients with confirmed cancer, proportion treated with stage I/II disease
Incidence of curative-intent treatment | From intervention start up to trial end at 1825 days
  Cumulative incidence (cases per standardized population) of initiation of curative-intent cancer treatment

SECONDARY OUTCOMES:
Cancer presenting as emergency | From date of cancer diagnosis to date of cancer treatment up to 7 days
  Among patients with confirmed cancer, proportion of cancer cases presenting as emergency (inpatient admission or death within 1 week of presentation with symptom).
Incident low probability cancer syndromes | Baseline
  Cumulative incidence (cases per standardized population) of presentation with low probability cancer syndromes
Final diagnosis within 8 weeks | From date of first clinic visit to date of cancer diagnosis or diagnosis excluding cancer, up to 56 days
  Among patients with moderate to high probability cancer symptoms, proportion with cancer diagnosis or exclusion of cancer diagnosis within 8 weeks of initial clinic visit
Incident invasive procedures in cancer suspects | From intervention start up to trial end at 1825 days
  Cumulative incidence (cases per standardized population) of presentation with low, moderate, or high probability cancer syndromes
Patients treated for cancer | From date of cancer diagnosis to date of cancer treatment up to 365 days
  Among patients with confirmed cancer, proportion of cancer cases receiving any cancer-specific therapy

CONTACTS AND LOCATIONS:
Overall Officials: Scott Dryden-Peterson, MD, MSc, Principal Investigator — Brigham and Women's Hospital, Botswana Harvard AIDS Institute
Locations (1):
- Botswana Harvard AIDS Institute, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: Yes
Data documentation and any de-identified information arising from this project will be deposited for sharing within the collaboration at a central secure, password protected electronic database managed initially by Botswana Harvard AIDS Institute with longer-term plans to move the database and responsibility for managing it to University of Botswana.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Following publication of primary study endpoints and for up to 5 years.
Access Criteria: IRB-approved (approval by Botswana Ministry of Health and Wellness required), cancer-related analyses consistent with informed consent document.

DOCUMENTS (1):
  • Informed Consent Form (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT04141449/ICF_000.pdf